CLINICAL TRIAL: NCT01312714
Title: A Randomized, Placebo-Controlled, Double Blind Study Evaluating the Effect of Cholecalciferol on Vasoactive Hormones, Heart Function, Arterial Stiffness, and Blood Pressure in Dialysis Patients.
Brief Title: Vitamin D3 Supplementation in Dialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, DMSc, Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBP-TL-2011
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: End-Stage Renal Disease
Keywords: Hemodialysis; Peritoneal dialysis; Vitamin D Deficiency; blood pressure; arterial stiffness; Heart function; Renin-angiotensin system; Calcium; FGF-23; Brain natriuretic peptide
MeSH Terms: conditions — Kidney Failure, Chronic; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Active Comparator)
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — 3 tablets of 1000 IU daily for 26 weeks
  Other Names: Vitamin D3
  Arms: Cholecalciferol
Drug: Placebo — 3 tablets of 1000 IU daily for 26 weeks
  Arms: Placebo

SUMMARY:
Vitamin D deficiency is highly prevalent among dialysis patients, and has been associated with cardiovascular risk factors such as increased aortic pulse wave velocity, blood pressure, inflammation, and brain natriuretic peptide. This study will evaluate the effect of 26 weeks of vitamin D3 supplementation in patients with end stage renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis or peritoneal dialysis > 3 months

Exclusion Criteria:

* Hypercalceamia
* Cancer
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of NT-proBNP | 26 weeks

SECONDARY OUTCOMES:
Plasma concentration of ionized calcium | 4 weeks
Plasma concentration of phosphate | 4 weeks
Plasma concentration of PTH | 4 weeks
Plasma concentration of 25-hydroxycholecalciferol | 4 weeks
24-hour blood pressure | 26 weeks
Plasma renin concentration | 26 weeks
Plasma concentration of angiotensin II | 26 weeks
Plasma concentration of aldosterone | 26 weeks
Arterial stiffness | 26 weeks
Serum concentration of FGF-23 | 26 weeks
Plasma concentration of AVP | 26 weeks
Plasma concentration of ANP | 26 weeks
Plasma concentration of TNF alpha | 26 weeks
Heart Function | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, M.D., M.Sci., Principal Investigator — Departments of Medical Research and Medicine
Locations (1):
- Departments of Medical Research and Medicine, Holstebro Hospital, Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Mose FH, Vase H, Larsen T, Kancir AS, Kosierkiewic R, Jonczy B, Hansen AB, Oczachowska-Kulik AE, Thomsen IM, Bech JN, Pedersen EB. Cardiovascular effects of cholecalciferol treatment in dialysis patients--a randomized controlled trial. BMC Nephrol. 2014 Mar 24;15:50. doi: 10.1186/1471-2369-15-50. PMID 24661355